CLINICAL TRIAL: NCT02795676
Title: A Randomized, Double Blind, Active Control Study of the Safety and Efficacy of PRX-102 Compared to Agalsidase Beta on Renal Function in Patients With Fabry Disease Previously Treated With Agalsidase Beta
Brief Title: Study of the Safety and Efficacy of PRX-102 Compared to Agalsidase Beta on Renal Function
Acronym: BALANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protalix (Industry)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB-102-F20
Record Dates: First submitted 2016-06-02; First posted 2016-06-10 (Estimated); Results first posted 2023-08-02 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Fabry Disease
Keywords: Glomerular filtration rate; Proteinuria; PRX-102; pegunigalsidase alfa; Fabry Disease
MeSH Terms: conditions — Fabry Disease; Proteinuria | interventions — agalsidase beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRX-102 (pegunigalsidase alfa) (Experimental): PRX-102 infusion every 2 weeks
  Interventions: Biological: PRX-102 (pegunigalsidase alfa)
- agalsidase beta (Active Comparator): agalsidase beta infusion every 2 weeks
  Interventions: Biological: agalsidase beta

INTERVENTIONS:
Biological: PRX-102 (pegunigalsidase alfa) — PRX-102 1 mg/kg every 2 weeks
  Other Names: pegunigalsidase alfa; Recombinant human alpha galactosidase-A
  Arms: PRX-102 (pegunigalsidase alfa)
Biological: agalsidase beta — agalsidase beta 1 mg/kg every 2 weeks
  Other Names: Fabrazyme
  Arms: agalsidase beta

SUMMARY:
This was a randomized, double-blind, active control study of the enzyme replacement therapy (ERT) drug PRX-102 (pegunigalsidase alfa) in Fabry disease patients with impaired renal function. Patients who had been treated for approximately 1 year with agalsidase beta and who had been on a stable dose of that product for at least 6 months were randomized in a 2:1 ratio to either switch to PRX-102 or to continue treatment with agalsidase beta. Both treatments were delivered by intravenous infusions every two weeks, at a dosage of 1 mg/kg.

DETAILED DESCRIPTION:
This was a randomized, double-blind, active control study examining the safety and efficacy of pegunigalsidase alfa (PRX-102) in Fabry disease patients with impaired renal function. Participants had to have been taking the licensed ERT drug agalsidase beta (Fabrazyme®) for at least 1 year prior to study entry, and to have been on a stable dose of that product for at least the last 6 months. Since the disease expresses itself differently in males and females, gender could have an impact on the therapeutic effect; thus, there was additionally a requirement that no more than 50% of the patients could be female.

Following screening, eligible patients were randomized in a 2:1 ratio to either switch to PRX-102 or continue treatment with agalsidase beta, with randomization stratified according to whether the urine protein-to-creatinine ratio (UPCR), a measure of kidney function, was above or below a specified threshold. Both products were administered as an intravenous infusion every 2 weeks, at a dosage of 1 mg/kg, for up to 24 months. Both patients and study staff were blinded as to which treatment was being given.

Patients who completed the study were invited to continue in a long-term open-label extension study, PB-102-F60, in which all participants would receive PRX-102 1 mg/kg every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic adult Fabry disease patients, age 18-60 years

  1. Males: Plasma and/or leucocyte alpha galactosidase activity (by activity assay) less than 30% mean normal levels and one or more of the characteristic features of Fabry disease

     i. neuropathic pain

     ii. cornea verticillata

     iii. clustered angiokeratoma
  2. Females:

     a. historical genetic test results consistent with Fabry pathogenic mutation and one or more of the described characteristic features of Fabry disease:

     i. neuropathic pain

     ii. cornea verticillata

     iii. clustered angiokeratoma

     b. or in the case of novel mutations a first degree male family member with Fabry disease with the same mutation, and one or more of the characteristic features of Fabry disease

     i. neuropathic pain

     ii. cornea verticillata

     iii. clustered angiokeratoma
* Screening eGFR by CKD-EPI equation 40 to 120 mL/min/1.73 m²
* Linear negative slope of eGFR based on at least 3 serum creatinine values over approximately 1 year (range of 9 to 18 months, including the value obtained at the screening visit) of ≥ 2 mL/min/1.73 m²/year
* Treatment with a dose of 1 mg/kg agalsidase beta per infusion every 2 weeks for at least one year and at least 80% of 13 (10.4) mg/kg total dose over the last 6 months.
* Female patients and male patients whose co-partners are of child-bearing potential agree to use a medically accepted method of contraception, not including the rhythm method.

Exclusion Criteria:

* History of anaphylaxis or Type 1 hypersensitivity reaction to agalsidase beta
* Known non-pathogenic Fabry mutations
* History of renal dialysis or transplantation
* History of acute kidney injury in the 12 months prior to screening, including specific kidney diseases (e.g., acute interstitial nephritis, acute glomerular and vasculitic renal diseases); non-specific conditions (e.g, ischemia, toxic injury); as well as extrarenal pathology (e.g., prerenal azotemia, and acute postrenal obstructive nephropathy)
* Angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) therapy initiated or dose changed in the 4 weeks prior to screening
* Patient with a screening eGFR value between 91-120 mL/min/1.73 m², having an historical eGFR value higher than 120 mL/min/1.73 m² (during 9 to 18 months before screening)
* Urine protein to creatinine ratio (UPCR) > 0.5 g/g and not treated with an ACE inhibitor or ARB
* Cardiovascular event (myocardial infarction, unstable angina) in the 6 month period before randomization
* Congestive heart failure NYHA Class IV
* Cerebrovascular event (stroke, transient ischemic attack) in the 6 month period before randomization
* Known history of hypersensitivity to Gadolinium contrast agent that is not managed by the use of pre-medication
* Female subjects who are pregnant, planning to become pregnant during the study, or are breastfeeding
* Presence of any medical, emotional, behavioral or psychological condition that, in the judgment of the Investigator and/or Medical Director, would interfere with the patient's compliance with the requirements of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (15):
  - UAB Medicine, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California Irvine Center, Orange, California
  - University of California San Diego, San Diego, California
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Iowa Hosptials and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Infusion Associates, Grand Rapids, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Institute of Metabolic Disease, Baylor Healthcare, Dallas, Texas
  - Renal Disease Research Institute, LLC - Dallas, Dallas, Texas
  - Eccles Primary Children's Outpatient Services Building, Salt Lake City, Utah
  - O+O Alpan LLC, Fairfax, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Vseobecna fakultni nemocnice v Praze, Prague, Czech Republic, Czechia
- Turku University Central Hospital, Turku, Finland
- Hôpital Raymond Poincaré, Paris, France
- Semmelweis Egyetem, Budapest, Hungary
- Azienda Ospedaliera Universitaria "Federico II", Napoli, Italy
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Haukeland University Hospital Klinisk Forskningspost, Bergen, Norway
- General Hospital Slovenj Gradec, Slovenj Gradec, Slovenia
- Hospital de Dia Quiron Zaragoza, Zaragoza, Spain
- Klinik und Poliklinik für Innere Medizin UniversitätsSpital Zürich, Zurich, Switzerland
- United Kingdom (4):
  - Institute of Metabolism and Systems Research, Edgbaston, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - The Royal Free Hospital, London
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azimpour K, Dorling P, Koulinska I, Kunduri S, Lan Z, Poritz J, Tremblay G, Raad-Faherty A. Health State Utility Values in Fabry Disease: Insights from the Pegunigalsidase Alfa Clinical Trials. Adv Ther. 2025 Mar;42(3):1421-1434. doi: 10.1007/s12325-024-03095-2. Epub 2025 Jan 23. PMID 39847314
- [Derived] Wallace EL, Goker-Alpan O, Wilcox WR, Holida M, Bernat J, Longo N, Linhart A, Hughes DA, Hopkin RJ, Tondel C, Langeveld M, Giraldo P, Pisani A, Germain DP, Mehta A, Deegan PB, Molnar MJ, Ortiz D, Jovanovic A, Muriello M, Barshop BA, Kimonis V, Vujkovac B, Nowak A, Geberhiwot T, Kantola I, Knoll J, Waldek S, Nedd K, Karaa A, Brill-Almon E, Alon S, Chertkoff R, Rocco R, Sakov A, Warnock DG. Head-to-head trial of pegunigalsidase alfa versus agalsidase beta in patients with Fabry disease and deteriorating renal function: results from the 2-year randomised phase III BALANCE study. J Med Genet. 2024 May 21;61(6):520-530. doi: 10.1136/jmg-2023-109445. PMID 37940383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Symptomatic adult Fabry patients who had been taking agalsidase beta for at least 1 year and on a stable dose for at least 6 months. No more than 50% could be female. Screening eGFR (CKD-EPI) 40 to 120 mL/min/1.73 m^2; Screening linear eGFR slope more negative than -2 mL/min/1.73 m^2/year based on at least 3 values over ~1 year.
Pre-assignment Details: Of the 78 randomized patients, 53 were assigned to the PRX-102 arm and 25 to the agalsidase beta arm. One PRX-102 patient withdrew consent before receiving the study product; accordingly, 77 patients were treated, 52 in the PRX-102 arm and 25 in the agalsidase beta arm.
Groups:
- PRX-102 (Pegunigalsidase Alfa): Pegunigalsidase alfa administered as an intravenous infusion every 2 weeks, at a dosage of 1 mg/kg
- Agalsidase Beta: Agalsidase beta administered as an intravenous infusion every 2 weeks, at a dosage of 1 mg/kg
Period: Overall Study
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta
Started | 53 | 25
Treated (One patient from PRX-102 arm withdrew consent before receiving the study product) | 52 | 25
Completed | 48 | 24
Not Completed | 5 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta | Total
Number analyzed (Participants) | 52 | 25 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 25 | 77
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (10.2) | 45.2 (9.6) | 44.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 7 | 30
  Male | 29 | 18 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 49 | 23 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 4 | 1 | 5
  Hungary | 0 | 1 | 1
  United States | 33 | 18 | 51
  Czechia | 1 | 0 | 1
  Norway | 1 | 1 | 2
  Finland | 0 | 1 | 1
  Italy | 2 | 1 | 3
  United Kingdom | 4 | 1 | 5
  Slovenia | 2 | 0 | 2
  France | 3 | 0 | 3
  Spain | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Annualized Change (Slope) in Estimated Glomerular Filtration Rate (eGFR)
Description: The individual annualized mean change (slope) in eGFR (mL/min/1.73 m^2/year) is an estimate of the individual patient's annualized change in eGFR, which is derived from the eGFR assessments over time, for up to 24 months.
  The individual annualized mean change (slope) in eGFR is estimated for each patient with at least 4 eGFR observations. For patients with fewer than 4 eGFR observations, the slope will be missing.
Time Frame: 24 months
Population: The Intent to Treat (ITT) population includes all randomized patients who received at least one dose of the assigned study medication with at least 4 eGFR observations.
  For 1 patient with fewer than 4 eGFR observations, the slope was missing.
Measure: Median (95% Confidence Interval); unit: mL/min/1.73 m^2/year
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta
Number analyzed (Participants) | 51 | 25
mL/min/1.73 m^2/year | -2.514 [-3.788 to -1.240] | -2.155 [-3.805 to -0.505]
Statistical Analysis 1: Comparison: PRX-102 (Pegunigalsidase Alfa) vs Agalsidase Beta; Test type: Non-Inferiority — Non-inferiority was to be declared if the lower bound of the confidence interval for the treatment difference is above the non-inferiority margin, which was met. No p-value was calculated as this is not relevant for non-inferiority; Regression, Linear; The primary efficacy analysis compared eGFR slope between the treatment arms using a 2-stage model with quantile regression; Median Difference (Final Values) = -0.359, 95% CI 2-sided [-2.444 to 1.726]

2. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR was calculated based on measured serum creatinine levels according to the CKD-EPI formula. The median values obtained at baseline and at Month 24 are reported.
  The change in eGFR from baseline measurement prior to first infusion to last measurement at Month 24 was summarized using descriptive statistics.
  The change was calculated for each subject and the reported value is the median (full range) of these changes.
Time Frame: Baseline and Month 24
Population: The Intent to Treat (ITT) population includes all randomized patients who received at least one dose of the assigned study medication.
Measure: Median (Full Range); unit: mL/min/1.73 m^2
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta
Number analyzed (Participants) | 52 | 25
mL/min/1.73 m^2
  Baseline | 73.45 [30.2 to 125.9] | 74.85 [34.1 to 107.6]
  Month 24 | 69.35 [27.6 to 113.7] | 74.48 [24.4 to 114.8]
  Change from Baseline to Month 24 | -2.39 [-36.9 to 21.8] | -3.20 [-18.0 to 16.8]

3. Secondary Outcome: Plasma Lyso-Gb3
Description: Globotriaosylsphingosine (lyso-Gb3) is a Fabry disease-specific biomarker measured in the plasma. The median concentrations obtained at baseline and at Month 24, and the change from baseline to Month 24 in median concentration, are reported.
  The change in Lyso-Gb3 from baseline measurement prior to first infusion to last measurement at Month 24 was summarized using descriptive statistics.
  The change was calculated for each subject and the reported value is the median (full range) of these changes.
Time Frame: Baseline and Month 24
Population: as for outcome 2
Measure: Median (Full Range); unit: nM
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta
Number analyzed (Participants) | 52 | 25
nM
  Baseline | 15.20 [0.8 to 143.9] | 17.60 [2.1 to 142.0]
  Month 24 | 18.80 [2.4 to 139.4] | 15.30 [1.5 to 71.2]
  Change from Baseline to Month 24 | 1.15 [-32.2 to 32.7] | -1.50 [-102.3 to 2.4]

4. Secondary Outcome: Short Form Brief Pain Inventory (BPI)
Description: The Short Form Brief Pain Inventory ( BPI) questioner is self-completed by patients regarding pain severity and interference.
  Descriptive statistics summarize the findings for the change from baseline at Week 104 for "Pain at Its Worst in Last 24 Hours".
  The severity of various aspects of pain scored on a scale of 0 to 10 ( no pain / pain as bad as you can imagine).
  The change in BPI from baseline measurement prior to first infusion to the last measurement at Month 24 was summarized using descriptive statistics.
  The change was calculated for each subject and the reported value is the mean (Standard Error) of these changes.
Time Frame: Baseline and Month 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta
Number analyzed (Participants) | 52 | 25
score on a scale
  Baseline | 3.5 (0.4) | 2.6 (0.6)
  Month 24 | 3.3 (0.5) | 3.0 (0.7)
  Change from Baseline to Month 24 | -0.1 (0.5) | 0.6 (0.6)

5. Secondary Outcome: Mainz Severity Score Index (MSSI)
Description: The Mainz Severity Score Index (MSSI) is an instrument that is specifically designed to measure the severity of Fabry disease signs/symptoms and to monitor the clinical course of the disease. The MSSI is administered by the investigator, and yields scores for general, neurological, cardiovascular, renal, and overall assessments. The overall score range from 0 to 76. An overall score of less than 20 points is considered mild signs and symptoms of Fabry disease, 20 to 40 is considered moderate, and greater than 40 is considered severe.
  The change in overall MSSI score from baseline measurement prior to first infusion to the last measurement at Month 24 was summarized using descriptive statistics.
  The change was calculated for each subject and the reported value is the mean (Standard Error) of these changes.
Time Frame: Baseline and Month 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta
Number analyzed (Participants) | 52 | 25
score on a scale
  Baseline | 23.18 (1.42) | 25.16 (2.14)
  Month 24 | 22.11 (1.80) | 27.09 (2.30)
  Change from Baseline to Month 24 | -2.07 (0.77) | 2.04 (1.10)

6. Secondary Outcome: Urine Protein/Creatinine Ratio (UPCR)
Description: The UPCR provides an estimate of protein excretion in urine, and is used as an indicator of the extent of chronic kidney disease. It was classified into three categories: 1) UPCR ≤ 0.5 gr/gr, 2) 0.5 gr/gr < UPCR < 1 gr/gr, 3) 1 gr/gr ≤ UPCR. The results are presented as the percentage of patients (%) in each category at baseline and Month 24.
  There are no statistical analyses for this endpoint.
Time Frame: Baseline and Month 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta
Number analyzed (Participants) | 52 | 25
percentage of participants
  UPCR ≤ 0.5 gr/gr, Baseline | 69 | 80
  UPCR ≤ 0.5 gr/gr, Month 24 | 76 | 75
  0.5 < UPCR < 1 gr/gr, Baseline | 17 | 8
  0.5 < UPCR < 1 gr/gr, Month 24 | 11 | 8
  UPCR ≥ 1 gr/gr, Baseline | 14 | 12
  UPCR ≥ 1 gr/gr, Month 24 | 13 | 17

7. Secondary Outcome: Left Ventricular Mass Index With Hypertrophy at Baseline
Description: Left Ventricular Mass Index (LVMI) based on cardiac MRI for patients with hypertrophy at baseline (for males, hypertrophy is above 91 g/m^2 and for females, above 77 g/m^2).
  The change in LVMI from baseline measurement prior to first infusion to the last measurement at Month 24 was summarized using descriptive statistics.
  The change was calculated for each subject and the reported value is the median (full range) of these changes.
Time Frame: Baseline and Month 24
Population: The Intent to Treat (ITT) population includes all randomized patients who received at least one dose of the assigned study medication.
  This analysis included the subset of patients in each treatment arm who had hypertrophy at baseline.
Measure: Median (Full Range); unit: g/m^2
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta
Number analyzed (Participants) | 12 | 9
g/m^2
  Baseline | 108.005 [81.77 to 168.42] | 103.030 [78.91 to 147.33]
  Month 24 | 118.130 [87.78 to 150.67] | 121.380 [63.78 to 187.23]
  Change from Baseline to Month 24 | -4.790 [-24.42 to 21.55] | 4.120 [-28.41 to 41.10]

8. Secondary Outcome: Left Ventricular Mass Index Without Hypertrophy at Baseline
Description: Left Ventricular Mass Index (LVMI) based on cardiac MRI for patients without hypertrophy at baseline (for males, hypertrophy is above 91 g/m^2 and for females, above 77 g/m^2).
  The change in LVMI from baseline measurement prior to first infusion to the last measurement at Month 24 was summarized using descriptive statistics.
  The change was calculated for each subject and the reported value is the median (full range) of these changes.
Time Frame: Baseline and Month 24
Population: The Intent to Treat (ITT) population includes all randomized patients who received at least one dose of the assigned study medication.
  This analysis included the subset of patients in each treatment arm who did not have hypertrophy at baseline.
Measure: Median (Full Range); unit: g/m^2
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta
Number analyzed (Participants) | 28 | 13
g/m^2
  Baseline | 55.555 [33.81 to 89.24] | 66.040 [35.74 to 86.92]
  Month 24 | 52.160 [35.80 to 100.01] | 62.520 [35.38 to 88.48]
  Change from Baseline to Month 24 | 1.990 [-29.37 to 18.37] | 0.515 [-13.69 to 11.15]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | PRX-102 (Pegunigalsidase Alfa) | Agalsidase Beta
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/25
Serious Adverse Events (participants affected / at risk) | 8/52 | 6/25
Other Adverse Events (participants affected / at risk) | 47/52 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRX-102 (Pegunigalsidase Alfa) (N=52) | Agalsidase Beta (N=25)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Medical device battery replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRX-102 (Pegunigalsidase Alfa) (N=52) | Agalsidase Beta (N=25)
Hypertension (Vascular disorders) | 3 (4) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 9 (10) | 4 (6)
Pyrexia (General disorders) | 5 (5) | 3 (4)
Oedema peripheral (General disorders) | 4 (9) | 3 (3)
Infusion site extravasation (General disorders) | 3 (4) | 0 (0)
Pain (General disorders) | 2 (3) | 3 (5)
Chest pain (General disorders) | 1 (1) | 3 (3)
Influenza like illness (General disorders) | 1 (1) | 3 (4)
Malaise (General disorders) | 1 (1) | 2 (3)
Chest discomfort (General disorders) | 0 (0) | 2 (3)
Seasonal allergy (Immune system disorders) | 4 (5) | 1 (2)
Hypersensitivity (Immune system disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (7)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Device occlusion (Product Issues) | 0 (0) | 2 (2)
Urine protein/creatinine ratio increased (Investigations) | 3 (5) | 0 (0)
Blood creatine increased (Investigations) | 2 (5) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (4)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 1 (3)
Palpitations (Cardiac disorders) | 3 (4) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 11 (19) | 5 (9)
Dizziness (Nervous system disorders) | 6 (8) | 2 (2)
Neuralgia (Nervous system disorders) | 4 (5) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0)
Sciatica (Nervous system disorders) | 3 (5) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 4 (8)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (15) | 6 (10)
Nausea (Gastrointestinal disorders) | 9 (10) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (8) | 3 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (7)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (3)
dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (23)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 6 (7) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (12) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (15) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Nasopharyngitis (Infections and infestations) | 11 (21) | 4 (6)
Sinusitis (Infections and infestations) | 8 (9) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 6 (12) | 4 (7)
Urinary tract infection (Infections and infestations) | 6 (6) | 3 (4)
Bronchitis (Infections and infestations) | 5 (6) | 5 (7)
Respiratory tract infection (Infections and infestations) | 3 (4) | 1 (3)
Viral infection (Infections and infestations) | 3 (3) | 3 (5)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 2 (4)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
* Small sample size
* Randomization of 2:1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT02795676/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT02795676/SAP_001.pdf